CLINICAL TRIAL: NCT02168426
Title: Randomized Control Trial on Seprafilm and Guardix in Preventing Ileus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Won-Suk Lee, Won-Suk Lee, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GDIRB2013-15
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Patient Under Going Colorectal and Stomach Cancer Surgery
MeSH Terms: interventions — guardix; Seprafilm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guardix (Active Comparator): 6g per body
  Interventions: Procedure: Guardix; Procedure: Seprafilm
- Seprafilm (Active Comparator): 1 sheet per body
  Interventions: Procedure: Guardix; Procedure: Seprafilm

INTERVENTIONS:
Procedure: Guardix — Applying 6g of guardix during abdominal surgery
  Other Names: Guardix, Sami pharmaceutical company; Seprafilm
Procedure: Seprafilm — Applying 1 sheet of seprafilm during abdominal surgery

SUMMARY:
The purpose of the study is to evaluate the efficacy of Seprafilm and guardix in reducing the incidence of bowel obstruction and to evaluate the incidence of all serious adverse events (SAEs) associated with the use of Seprafilm and guardix occurring within 30 days postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of GI cancer
* Operable

Exclusion Criteria:

* Withdrew consent
* Pregnant
* Ascites
* Distant metastasis
* Liver dysfunction (serum total bilirubin >2.0 mg/dL)
* Renal failure (serum creatinine >1.5 mg/dL)
* A past history of small bowel obstruction.

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
ileus rate | within 60 days
  Reducing the incidence of bowel obstruction following intestinal resection, and subsequently, reducing the number of re-operations

SECONDARY OUTCOMES:
adverse effect rate | within 60 days

CONTACTS AND LOCATIONS:
Locations (1):
- Won-Suk Lee, Incheon, South Korea